CLINICAL TRIAL: NCT04008628
Title: Analgesia by 50%/50% Nitrous Oxide/Oxygen Mixture for Nasogastric Catheterization in Children Aged 3 Months to 3 Years
Brief Title: Nitrous Oxide for Analgesia During Nasogastric Tube Placement in Young Children
Acronym: SONGER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHRIP18164
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Mild to Moderate Dehydration
Keywords: Pain; nasogastric tube; children; infants; analgesia; nitrous oxide
MeSH Terms: conditions — Pain; Agnosia | interventions — Nitrous Oxide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The primary outcome will be assessed on video recordings of the procedures which will be prepared so that assessors will not know to which group the children assigned. This correspond to a blind assessment of the primary outcome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nitrous oxide (Active Comparator): Inhalation of a 50%/50% mixture of nitrous oxide and oxygen. Reassurance of the child during procedure
  Interventions: Drug: Nitrous Oxide
- Standard care (No Intervention): Infants will be reassured as currently performed in routine clinical practice

INTERVENTIONS:
Drug: Nitrous Oxide — Inhalation of a 50%/50% nitrous oxide/oxygen mixture (Kalinox®)
  Arms: Nitrous oxide

SUMMARY:
Since nitrous oxide/oxygen mixture is effective to reduce pain and anxiety induced by various painful procedures in children, the investigators hypothesized that its inhalation would reduce pain during nasogastric tube placement in young children.

The purpose of this study is to evaluate the analgesic efficacy of 50%/50% nitrous/oxide mixture in reducing pain induced by nasogastric tube insertion in children aged 3 months to 3 years in the pediatric emergency department.

DETAILED DESCRIPTION:
In the context of mild to moderate dehydration in young children, enteral rehydration is the treatment of choice because it is more physiological than parenteral rehydration which has more serious side effects. Thus, nasogastric tube placement has become a more common procedure in the pediatric emergency care setting. Although, it is widely accepted that this procedure is invasive and painful, to date, no analgesic approach has been shown to be effective for children aged 3 months to 3 years. Currently, standard care is the placement of nasogastric tube without any analgesic intervention.

Inhalation of nitrous oxide mixed with oxygen (50/50) has been shown to be effective to reduce pain and anxiety induced by invasive procedures in children, adolescents and adults. Its use is very safe and it is associated with only minor and transient side effects such as nausea, vomiting or dizziness in les than 10% of patients. Its use is very common in many countries such as France, United Kingdom, The Netherlands or Australia. The investigators hypothesized that its inhalation would reduce pain during nasogastric tube placement in young children.

The purpose of this study is to evaluate the analgesic efficacy of 50%/50% nitrous/oxide mixture in reducing pain induced by nasogastric tube insertion in children aged 3 months to 3 years in the pediatric emergency department.

A randomized controlled trial will be performed in two pediatric emergency departments to assess the efficacy of 50/50 nitrous oxide/oxygen during nasogastric tube insertion. The control group will receive standard care.

Primary outcome: Pain assessed with the FLACC scale during tube insertion

The investigators believe that this randomized study comparing nitrous oxide inhalation against current practice (no analgesic means) will highlight the intensity of pain caused by nasogastric tube placement and will assess the effectiveness of nitrous oxide inhalation to reduce pain and anxiety induced by the procedure

ELIGIBILITY:
Inclusion Criteria:

* Child from 3 months to 3 years old.
* Admission to the Pediatric Emergency Department
* Medical prescription for the insertion of a nasogastric tube.
* Child with gastroenteritis and / or bronchiolitis and / or food intolerance with mild to moderate dehydration
* Parental presence and parental consent

Exclusion Criteria:

* Vital emergency.
* Refusal of parents.
* Refusal of parents to be filmed
* Child already included in the study or in course of participation in another study.
* Tube placement performed by a medical student or nursing student.
* Patient requiring 100% oxygen ventilation.
* No social security.
* Child with a mental handicap or known retardation
* History of child intolerance to Nitrous oxide ( excessive sedation or respiratory depression during previous use)
* Child with head trauma in the previous 3 days

Premature discontinuation of study participation :

* Parents' request to stop participating in the study.
* Insertion of the nasogastric tube is not possible

Ages: 3 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Pain during nasogastric tube insertion | From the beginning of the procedures until 2 minutes after final positioning of the tube
  Pain will be assessed during nasogastric tube insertion with the Face Legs Activity Cry Consolability (FLACC) scale composed of five scale (face, legs, activities, shouting, consolability). Each ranks from 0 to 2 : 0 is no pain, 1 is average pain, 2 is a strong pain The outcome measure is the sum of these five subscales: from 0 (better outcome) to 10 (worse outcome).

SECONDARY OUTCOMES:
Parent's anxiety 10 scale. | During procedure
  The parent evaluates himself his anxiety. It's a simple scale graduate one by one, from 0 (better outcome) to 10 (worse outcome). Based on their subjective interpretation of their own anxiety
Child's constraint needed during the procedure | During procedure
  Scale for grading the level of constraint during the procedure It is composed to three subscales from 0 to 3 (head, arms, legs). 0 is no contention, 1 is soft hold, 2 is firm support, 3 is very firm hold And one subscale from 0 to 1 (trunk). 0 is no contention, 1 is necessary maintenance.
  The outcome measure is the sum of these four subscales: from 0 (better outcome, that is to say no contention) to 10 (strongest contention).
The potential side effects of the mixture 50%/50% nitrous oxide/oxygen for a brief inhalation are : Euphoria, dreaming, hallucinations, sedation, headaches, nausea, and vomiting. | from the start of inhalation to nearly 5 to 10 minutes after the end of inhalation
  The rate of side effects will be described

CONTACTS AND LOCATIONS:
Overall Officials: Marie Beauchet-Filleau, nurse, Principal Investigator — Trousseau Hospital, pediatric emergency; Ricardo Carbajal, Professor, Study Director — Trousseau Hospital, pediatric emergency
Locations (4):
- France (4):
  - Ambroise Paré hospital, Pediatric emergency department, Boulogne-Billancourt
  - Louis Mourier Hospital, Pediatric emergency department, Colombes
  - Trousseau Hospital, Pediatric emergency department, Paris, Île-de-France Region
  - Poissy Hospital, Pediatric emergency department, Poissy, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No